CLINICAL TRIAL: NCT04648462
Title: Proton Therapy Research Infrastructure- ProTRAIT- Neuro-oncology
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University Medical Center Groningen (Other); HollandPTC (Industry); Erasmus Medical Center (Other); Leiden University Medical Center (Other); Medical Center Haaglanden (Other); Maastro Clinic, The Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: ProTRAIT-neuro
Record Dates: First submitted 2020-11-06; First posted 2020-12-01 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Astrocytoma; Ependymoma; Ganglioglioma; Oligodendroglioma; Optic Nerve Glioma; Meningioma; Nerve Sheath Neoplasms; Adenoma; Craniopharyngioma; Hemangiopericytoma; Germinoma; Neurilemmoma
MeSH Terms: conditions — Astrocytoma; Ependymoma; Ganglioglioma; Oligodendroglioma; Optic Nerve Glioma; Meningioma; Nerve Sheath Neoplasms; Adenoma; Craniopharyngioma; Hemangiopericytoma; Germinoma; Neurilemmoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ProTRAIT — The participants are seen at the outpatient clinic by a physician, physician assistant or trial nurse at standard follow-up times at 2.5, 5, 7.5 and 10 years after radiotherapy.

SUMMARY:
The first proton therapy treatments in the Netherlands have taken place in 2018. Due to the physical properties of protons, proton therapy has tremendous potential to reduce the radiation dose to the healthy, tumour-surrounding tissues. In turn, this leads to less radiation-induced complications, and a decrease in the formation of secondary tumours. The Netherlands has spearheaded the development of the model-based approach (MBA) for the selection of patients for proton therapy when applied to prevent radiation-induced complications. In MBA, a pre-treatment in-silico planning study is done, comparing proton and photon treatment plans in each individual patient, to determine (1) whether there is a significant difference in dose in the relevant organs at risk (ΔDose), and (2) whether this dose difference translates into an expected clinical benefit in terms of NormalTissue Complication Probabilities (ΔNTCP). To translate ΔDose into ΔNTCP, NTCP-models are used, which are prediction models describing the relation between dose parameters and the likelihood of radiation-induced complications. The Dutch Society for Radiotherapy and Oncology (NVRO) setup the selection criteria for proton therapy in 2015, taking into account toxicity and NTCP. However, NTCP-models can be affected by changes in the irradiation technique. Therefore, it is paramount to continuously update and validate these NTCP-models in subsequent patient cohorts treated with new techniques. In ProTRAIT, a Findable, Accessible, Interoperable and Reusable (FAIR)data infrastructure for both clinical and 3D image and 3D dose information has been developed and deployed for proton therapy in the Netherlands. It allows for a prospective, standardized, multi-centric data from all Dutch proton and a representative group of photon therapy patients.

ELIGIBILITY:
Inclusion Criteria:

1. All brain tumors with a favorable prognosis (median survival > 10 year)
2. Age ≥ 18 years
3. ECOG performance status 0 - 1 / Karnofsky performance status 80 - 100
4. No - minimal neurocognitive impairment
5. Dosimetrical gain of protontherapy relative to photontherapy (≥5% on supratentorial brain dose or hippocampi)
6. Informed consent

Exclusion Criteria:

1. Not eligible for chemotherapy
2. Eligible for stereotactic radiotherapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All neuro-oncological patients treated with proton therapy at one of the three proton centers in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive failure at 5 years | 5 years after radiotherapy
  Time to neurocognitive failure, defined as the time from last radiotherapeutic treatment to the first instance of a measured HVLT-dr of -1.5Z based on the normal data

SECONDARY OUTCOMES:
HVLT- delayed recall decline at 5 years | 5 years after radiotherapy
  HVLT- delayed recall decline of -1.5Z compared to baseline at 5 years, using the RCI method based on the normal data
HVLT total recall decline at 5 years | 5 years after radiotherapy
  HVLT total recall decline of -1.5Z compared to baseline at 5 years, using the RCI method based on the normal data
TMT a decline at 5 years | 5 years after radiotherapy
  TMT a decline of -1.5Z compared to baseline at 5 years, using the RCI method based on the normal data
TMT b decline at 5 years | 5 years after radiotherapy
  TMT b decline of -1.5Z compared to baseline at 5 years, using the RCI method based on the normal data
COWA total decline at 5 years | 5 years after radiotherapy
  COWA total decline of -1.5Z compared to baseline at 5 years, using the RCI method based on the normal data

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Eekers, Principal Investigator — Maastro Clinic, The Netherlands; Danielle Eekers, Study Chair — Maastro Clinic, The Netherlands; Hiske van der Weide, Principal Investigator — UMC Groningen; M Kramer, Principal Investigator — UMC Groningen; Yvonne Klaver, Principal Investigator — HollandPTC; M Kroesen, Principal Investigator — HollandPTC; A Mendez Romero, Principal Investigator — Erasmus Medical Center; J Jaspers, Principal Investigator — Erasmus Medical Center; I Coremans, Principal Investigator — Leiden University Medical Center; Jaap Zindler, Principal Investigator — Medical Center Haaglanden; Inge Compter, Principal Investigator — Maastro Clinic, The Netherlands
Locations (3):
- Netherlands (3):
  - Maastricht Radiation Oncology, Maastricht, Limburg
  - Holland PTC, Delft, South Holland
  - Universitair Medisch Centrum Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No